CLINICAL TRIAL: NCT05728658
Title: A Phase I Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Preliminary Efficacy of ICP-248 as Monotherapy or in Combination Therapy in Patients With Mature B-cell Malignancies
Brief Title: The Study of ICP-248 in Patients With Mature B-cell Malignancies
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Beijing InnoCare Pharma Tech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: ICP-CL-01201
Record Dates: First submitted 2023-01-12; First posted 2023-02-15 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Hematological Malignancies
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (7):
- Dose-Escalation Cohort - R/R CLL/SLL and R/R MCL (Experimental): ICP-248 was divided into 6 dose groups, and each dose group was given progressively
  Interventions: Drug: ICP-248
- Dose-Expansion Cohort A/B/C/D/E/F (R/R CLL/SLL、R/R MCL、R/R B-NHL) (Experimental): Participants will receive ICP-248 daily with a weekly ramp-up schedule from Cycle 1 day 1.
  Interventions: Drug: ICP-248
- Dose-Expansion Cohort G(R/R MCL) (Experimental): Participants will receive ICP-248 daily with a ramp-up phase, and will receive Orelabrutinib 150 mg daily, until progressive disease (PD),intolerable toxicity,withdrawal of consent, loss to follow-up, initiation of other anti-cancer therapy, death,or end of study,whichever occurs first.
  Interventions: Drug: ICP-248+Orelabrutinib
- Dose-Expansion Cohort H(R/R MZL) (Experimental): Participants will receive ICP-248 daily with a weekly ramp-up schedule and Orelabrutinib 150 mg daily from Cycle 1 day 1, until progressive disease (PD),intolerable toxicity,withdrawal of consent, loss to follow-up, initiation of other anti-cancer therapy, death,or end of study,whichever occurs first.
  Interventions: Drug: ICP-248+Orelabrutinib
- Dose-Expansion Cohort I(R/R CLL/SLL) (Experimental): Participants will receive ICP-248 daily with a weekly ramp-up schedule from Cycle 1 day 1, and will receive 375 mg/m2 Rituximab on day 1 of each cycle from C1 to C6,or until progressive disease (PD),intolerable toxicity,withdrawal of consent, loss to follow-up, initiation of other anti-cancer therapy, death,or end of study,whichever occurs first.
  Interventions: Drug: ICP-248 +Rituximab
- Dose-Expansion Cohort J(R/R CLL/SLL) (Experimental): Participants will receive Orelabrutinib 150 mg daily from cycle 1 day 1, and will receive ICP-248 daily with a daily ramp-up schedule from Cycle 3 day 1, until progressive disease (PD),intolerable toxicity,withdrawal of consent, loss to follow-up, initiation of other anti-cancer therapy, death,or end of study,whichever occurs first.
  Interventions: Drug: ICP-248+Orelabrutinib
- Dose-Expansion Cohort K(MCL) (Experimental): Participants will receive Orelabrutinib 150 mg daily from cycle 1 day 1, and Rituximab 375 mg per square meter was infused intravenously on day 1 of each cycle from C1-6 and on day 1 of every two cycles from C7D1 onwards, and ICP-248 daily with a weekly ramp-up schedule from cycle 3 day 1. The treatment will continue up to a maximum of 24 cycles, or until progressive disease (PD),intolerable toxicity,withdrawal of consent, loss to follow-up, initiation of other anti-cancer therapy, death,or end of study,whichever occurs first.
  Interventions: Drug: ICP-248+Orelabrutinib+Rituximab

INTERVENTIONS:
Drug: ICP-248 — Eligible patients will receive ICP-248 orally as per the protocol, once daily for every 28 days as one treatment cycle (except for the food effect investigation phase), until progressive disease (PD), intolerable toxicity, withdrawal of consent, loss to follow-up, initiation of other anti-cancer therapy, death, or end of study, whichever occurs first.
  Arms: Dose-Escalation Cohort - R/R CLL/SLL and R/R MCL
Drug: ICP-248 — Eligible patients will receive ICP-248 orally as specified in the treatment arm.
  Arms: Dose-Expansion Cohort A/B/C/D/E/F (R/R CLL/SLL、R/R MCL、R/R B-NHL)
Drug: ICP-248+Orelabrutinib — Eligible patients will receive ICP-248 and Orelabrutinib as specified in the treatment arm.
  Arms: Dose-Expansion Cohort G(R/R MCL)
Drug: ICP-248+Orelabrutinib — Eligible patients will receive ICP-248 and Orelabrutinib as specified in the treatment arm.
  Arms: Dose-Expansion Cohort H(R/R MZL)
Drug: ICP-248 +Rituximab — Eligible patients will receive ICP-248 and Rituximab as specified in the treatment arm.
  Arms: Dose-Expansion Cohort I(R/R CLL/SLL)
Drug: ICP-248+Orelabrutinib — Eligible patients will receive ICP-248 and Orelabrutinib as specified in the treatment arm.
  Arms: Dose-Expansion Cohort J(R/R CLL/SLL)
Drug: ICP-248+Orelabrutinib+Rituximab — Eligible patients will receive ICP-248 and Orelabrutinib and Rituximab as specified in the treatment arm.
  Arms: Dose-Expansion Cohort K(MCL)

SUMMARY:
A Phase I Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Preliminary Efficacy of ICP-248 as Monotherapy or in Combination Therapy in Patients with Mature B-cell Malignancies.This study consists of two parts: Part 1 dose-finding period and Part 2 dose expansion period.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 and ≤ 80 years.
2. One of the following histopathologically and/or flow cytometry-confirmed diseases according to the 2016 World Health Organization (WHO) classification criteria for lymphohematopoietic neoplasms or meeting the International Workshop on Chronic Lymphocytic Leukemia (iwCLL) criteria: Histopathologically and/or flow cytometry-confirmed CLL/SLL; Pathologically confirmed MCL; Pathologically confirmed B-NHL, including diffuse large B-cell lymphoma (DLBCL), follicular lymphoma (FL), marginal zone lymphoma (MZL), and lymphoplasmacytic lymphoma (LPL).
3. Relapsed disease or refractory disease
4. For subjects with B-NHL: Patients must have measurable diseasePatients with an Eastern Cooperative Oncology Group (ECOG) performance status (PS) score of ≤ 2 and a life expectancy of ≥ 6 months.
5. Adequate hematologic function.
6. Patients with basically normal coagulation function.
7. Patients with adequate hepatic, renal, pulmonary and cardiac functions.
8. CLL/SLL Patients with an absolute lymphocyte count ≥ 50 x 109/L and any lymph nodes ≥ 5 cm in the long diameter or CLL/SLL or B-NHL patients with any lymph nodes ≥ 10 cm in the long diameter will be enrolled in the study after weighing the risks and benefits with the sponsor's MM.
9. Female patients of childbearing potential must have a negative blood pregnancy test within 7 days prior to the first dose of the investigational product; patients of childbearing potential (males and females) must agree to use a reliable birth control method (hormonal or barrier method or abstinence) with their partners from signing the ICF until 90 days after the last dose.The last ICP- 248 dose or within one month after the last dose of Orelabrutinib Or within 12 months after the last dose of Rituximab (whichever is longer).
10. Subjects are able to communicate with the investigator well and to complete the study as specified in the study.
11. Before the trial, the subjects shall understand the nature, significance, possible benefits, inconveniences and potential risks, as well as the study procedures of the trial in detail and voluntarily sign the written Informed Consent Form (ICF).
12. Subjects with CLL/SLL must have an indication for treatment as judged by the investigator.

Exclusion Criteria:

1. Prior malignancy (other than the disease under study) within 2 years before study entryKnown
2. Central nervous system involvement by lymphoma/leukemia
3. Underlying medical conditions that, in the investigator's opinion, will render the administration of the investigational product hazardous or obscure the interpretation of the safety or efficacy results.
4. Prior autologous stem cell transplant (unless ≥ 3 months after transplant); or prior chimeric cell therapy (unless ≥ 3 months after cell infusion).
5. Received a BCL-2 inhibitor prior to initial use of the investigational drug and did not achieve disease remission or disease recurrence/progression on treatment; Disease recurrence/progression after stopping or ending BCL-2 inhibitor therapy is acceptable.
6. A history of allogeneic stem cell transplantation.
7. Anti-cancer therapy within 14 days prior to the first dose of the investigational product
8. An interval of less than 5 half-lives from the last dose of a strong CYP3A inhibitor or inducer (chemical agent, traditional Chinese medicine and dietary supplement) to the first dose of the investigational product, or a plan to use concurrently medications, dietary supplements or food (e.g., grapefruit or grapefruit juice) with strong CYP3A inhibitory or inductive effect during study participation.
9. Patients who have undergone major organ surgery (excluding aspiration biopsy) or significant trauma within 28 days prior to the first dose of the investigational product, or who require elective surgery during the trial.
10. Patients who have received a live attenuated vaccine within 28 days prior to the first dose of the investigational product (except for vaccination to prevent a major public health event).
11. Presence of active infection that currently requires intravenous systemic anti-infective therapy.
12. Patients with active hepatitis B or C virus infection.
13. History of immunodeficiency, including a positive human immunodeficiency virus (HIV) antibody test.
14. History of significant cardiovascular disease
15. Patients with previous or concomitant central nervous system disordersHistory or current evidence of severe interstitial lung disease.
16. ≥ Grade 2 toxicity due to prior anti-cancer therapy at enrollment (except for alopecia, ANC, hemoglobin and PLT). For ANC, hemoglobin and PLT, please follow the inclusion criteria.
17. History of severe bleeding disorder
18. Known alcohol or drug dependence.
19. Presence of mental disorders or poor compliance.
20. Female patients who are pregnant or lactating.
21. Unable to swallow tablets or disease significantly affecting gastrointestinal function.
22. Hypersensitivity to the active substance or excipients of ICP-248 tablets or Orelabrutinib tablets (only applicable to subjects in cohort G/H/J/K).Severe allergic reaction or intolerance to murine monoclonal antibodies or murine products.

23 Invasive mantle cell lymphoma, such as mother cell subtypes, polymorphic subtypes, or Ki-67 proliferation index>50%, must be discussed with the sponsor's medical monitor regarding patient benefits and risks before being included in this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 191 (Estimated)
Dates: Start 2023-03-09 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose and recommended Phase 2 dose | 5 years
  To evaluate the safety and tolerability of ICP-248 monotherapy or combination with Orelabrutinib in the selected B-cell malignancies and to determine the maximum tolerated dose (MTD) and recommended Phase 2 dose (RP2D) of ICP-248
To investigate the incidence, nature and severity of adverse events (AE) according to NCI-CTCAE V5.0 or iwCLL2018 evaluation criteria. | 5 years
To evaluate the investigator-assessed overall response rate (ORR) of ICP-248 monotherapy or combination therapy at the recommended phase II dose (RP2D) . | 5 years

SECONDARY OUTCOMES:
Pharmacokinetic (PK) profile - Area under curve (AUC0-t) | 5 years
  To evaluate the AUC0-t after single administration of ICP-248 and steady state of ICP-248.
Pharmacokinetic (PK) profile - Maximum Concentration (Cmax) | 5 years
  To evaluate the Cmax after single administration of ICP-248 and steady state of ICP-248.
Pharmacokinetic (PK) profile - Time to maximum concentration (Tmax) | 5 years
  To evaluate the Tmax after single administration of ICP-248 and steady state of ICP-248.
Pharmacokinetic (PK) profile - Apparent clearance (CL/F) | 5 years
  To evaluate the CL/F after single administration of ICP-248 and steady state of ICP-248.
Preliminary efficacy - Complete response rate (CRR) | 5 years
  To evaluate the preliminary efficacy of ICP-248 monotherapy in the evaluated disease types as measured by investigator-assessed complete response rate (CRR).
Preliminary efficacy - Progression-free survival (PFS) | 5 years
  To evaluate the preliminary efficacy of ICP-248 monotherapy in the evaluated disease types as measured by investigator-assessed progression-free survival (PFS).
Preliminary efficacy - Duration of response (DOR) | 5 years
  To evaluate the preliminary efficacy of ICP-248 monotherapy in the evaluated disease types as measured by investigator-assessed duration of response (DOR).
Preliminary efficacy - Overall survival (OS) | 5 years
  To evaluate the preliminary efficacy of ICP-248 monotherapy in the evaluated disease types as measured by investigator-assessed overall survival (OS).
AUC of ICP-248 under different feeding conditions | 5 years
  To evaluate the AUC of ICP-248 under different feeding conditions.
Maximum Concentration (Cmax) of ICP-248 under different feeding conditions | 5 years
  To evaluate the Cmax of ICP-248 under different feeding conditions.
Time to maximum concentration (Tmax) of ICP-248 under different feeding conditions | 5 years
  To evaluate the Tmax of ICP-248 under different feeding conditions.

CONTACTS AND LOCATIONS:
Locations (22):
- China (22):
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - The Central Hospital of Wuhan, Wuhan, Hubei
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Jiangxi Cancer Hospital, Nanchang, Jiangxi
  - The Second Hospital of Dalian Medical University, Dalian, Liaoning
  - Shenyang Hospital Of China Medical University, Shenyang, Liaoning
  - Shandong cancer hospital, Jinan, Shandong
  - Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Hematology Hospital, Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No